CLINICAL TRIAL: NCT04348786
Title: Comparing the Efficacy of 14-day Therapy Doxycycline With Bismuth Subsalicylate Versus Levofloxacin With Tinidazole on Rate of Eradication of Helicobacter Pylori Infected Patients on Syrian Population
Brief Title: Comparing Efficacy of 14-day Therapy Doxycycline With Bismuth Subsalicylate Versus Levofloxacin With Tinadizole on Treatment Helicobacter Pylori
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Damascus Hospital (Other)
Responsible Party: Principal Investigator, Marouf Alhalabi, head of digestive diseases department, Damascus Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G1-19
Record Dates: First submitted 2020-01-29; First posted 2020-04-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Helicobacter Pylori Infection
Keywords: Doxycyclien; Bismuth Subsalicylate; Helicobacter Pylori; levofloxacine; tinadizole
MeSH Terms: interventions — Doxycycline; Esomeprazole; bismuth subsalicylate; Levofloxacin; Amoxicillin; Omeprazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxycyclien (Experimental): Measure eradication rate of Helicobacter pylori infection with Doxycycline and bismuth subsalicylate
  Interventions: Drug: Doxycycline
- Levofloxacine (Active Comparator): Measure eradication rate of Helicobacter pylori infection with Livofloxacine and tinadizole
  Interventions: Drug: Levofloxacin 500mg

INTERVENTIONS:
Drug: Doxycycline — Doxycylcine 100 mg bid ,esomprazole 20 bid,Bismuth subsalicylate 262 tab.2 tab q.i.d,Tinadizole 500 bid
  Other Names: Tinadizole; Esomeprazole; Bismuth subsalicylate
  Arms: Doxycyclien
Drug: Levofloxacin 500mg — Levofloxacin 500 mg qd, amoxicillin 500 2cab bid,Tinadizole 500 bid, esomprazole 20 bid
  Other Names: Amoxicilline; Esomeprazol; Tinadiole
  Arms: Levofloxacine

SUMMARY:
Comparison Efficacy of 10-days Therapy with Doxycycline with Bismuth Subsalicylate Versus Levofloxacine with Tinadizole on Eradication of Helicobacter Pylori in Syrian population.

ELIGIBILITY:
Inclusion Criteria:

* Patients are aged greater than 18 years old who have H. pylori infection diagnosed by any of following three methods:
* Positive rapid urease test (CLOtest).
* Histologic evidence of H. pylori by modified Giemsa staining.
* Positive 13C-urea breath test. without prior eradication therapy and are willing to receive therapy.

Exclusion Criteria:

* Children and teenagers aged less than 18 years.
* Previous eradication treatment for H. pylori.
* Patients who took any drug, which could influence the study results such as proton pump inhibitor, H2 blocker, mucosal protective agent and antibiotics.
* History of gastrectomy.
* Gastric malignancy, including adenocarcinoma and lymphoma,
* Previous allergic reaction to antibiotics (Amoxicillin, Tinadizole,
* Doxycycline,Bismuth subsalicylate,) and prompt pump inhibitors (Es- omeprazole).
* Contraindication to treatment drugs.
* Pregnant or lactating women.
* Severe concurrent disease.
* Liver cirrhosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Eradication rate of Helicobacter pylori infection | 8 week from begning of treatment
  Eradication rate of Helicobacter infected patients

CONTACTS AND LOCATIONS:
Overall Officials: Marouf M Alhalabi, MD, Principal Investigator — general assambly of damascus hospital
Locations (1):
- General Assembly of Damascus Hospital, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: Within 5 year of study completion

REFERENCES:
- [Derived] Alhalabi M, Alassi MW, Alaa Eddin K, Cheha K. Efficacy of two-week therapy with doxycycline-based quadruple regimen versus levofloxacin concomitant regimen for helicobacter pylori infection: a prospective single-center randomized controlled trial. BMC Infect Dis. 2021 Jul 4;21(1):642. doi: 10.1186/s12879-021-06356-5. PMID 34218802